CLINICAL TRIAL: NCT01507688
Title: Stroke Self-Management: Effect on Function and Stroke Quality of Life
Brief Title: Stroke Self-Management: Effect on Function and Stroke Specific Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SDP 10-379
Record Dates: First submitted 2012-01-04; First posted 2012-01-11 (Estimated); Results first posted 2019-04-01 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Stroke
Keywords: Stroke; Self-Management; Transient ischemic attack; Self-Efficacy
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 SSM Intervention (Experimental): Stroke self-management program- Participants randomized to this program will receive 6 bi-weekly telephone sessions during the first 3 months followed by 3 monthly reinforcement telephone sessions coupled with 3 monthly group sessions during months 4-6.
  Interventions: Behavioral: Stroke Self-Management
- Arm 2 Usual Care (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Stroke Self-Management — Stroke self-management program- Participants randomized to this program will receive 6 bi-weekly telephone sessions during the first 3 months followed by 3 monthly reinforcement telephone sessions coupled with 3 monthly group sessions during months 4-6.
  Arms: Arm 1 SSM Intervention

SUMMARY:
The experience of a stroke event may result in a disruption to the survivor's daily life. Patients with stroke have reported fears of permanent disability and major concerns over their ability to recover and be productive and engaged with family, friends and coworkers. To enhance recovery from stroke, the investigators designed a stroke self-management program and have pilot tested the program among Veterans recovering from stroke/TIA. The study is a three-site, randomized controlled trial designed to test the efficacy of a stroke self-management program. The intervention program includes 6 bi-weekly sessions over months 1-3 followed by monthly telephone calls as the investigators administered in the investigators' pilot study during months 4-6 for a total length of program duration of 6 months. The investigators have added 3 monthly group support sessions during months 4-6 for additional peer support. Thus, participants will receive bi-monthly support during months 4-6. The three intervention sites include the Jesse Brown VAMC in Chicago, the Roudebush VAMC in Indianapolis, and the IU Health Methodist Hospital in Indianapolis, Indiana. The three hospitals represent facilities with a small, moderate, and large volume of acute stroke care, respectively. Additionally, Methodist Hospital includes a greater proportion of women which enables us to study the patterns and preferences of women with stroke/TIA and tailor the investigators' future programs to prepare for the increasing female Veteran population.

DETAILED DESCRIPTION:
Stroke Self-Management: Effect on Function and Stroke Quality of Life Anticipated Impacts on Participant's Healthcare: This planned evaluation of the investigators' stroke self-management program may improve the patient's healthcare by establishing an evidence-based program for which VA case managers may implement to improve patient self-management and the health-related quality of life of stroke survivors. This program produced standardized manuals for case managers and stroke survivors that may be used in the field, in the patient medical care home and via telehealth.

Project Background: Stroke is prevalent and associated with increased morbidity and mortality. Stroke is the leading cause of long-term disability in the US. Within the VA, approximately 60,000 patients had a primary outpatient encounter for stroke during fiscal year 2010 (FY10). Data from the Office of Quality and Performance (OQP) Stroke Special Study demonstrate that more than 5,000 Veterans were admitted to a VA facility for acute ischemic stroke in FY07 and another 5000 Veterans with a transient ischemic attack (TIA) or mini-stroke, were admitted in a VA facility or received care at an urgent clinic or emergency department in VA. The total VA cost of stroke treatment was almost $315 million in FY05, with a cost per patient of over $18,000. Stroke/TIA survivors are at elevated risk for future vascular events and yet, there are no systematic post stroke programs offered widely in VA designed to reduce this risk and increase stroke specific quality of life in Veterans. The investigators recently developed and pilot tested a stroke self-management program that adapted the Stanford Chronic Disease program for stroke.

Project Objectives: The objectives of this project were to: 1. Conduct a randomized trial comparing stroke survivors randomly assigned to receive a stroke self-management program on patient functioning, stroke self-management, and stroke specific quality of life compared to stroke survivors assigned to usual care; and 2. Conduct a summative evaluation among VA clinical providers, patients with stroke and their caregivers to understand the barriers and facilitators of implementing the stroke self-management program.

Project Methods: To accomplish these aims, the investigators employed mixed methods. For the first aim, the investigators conducted a randomized controlled trial comparing subjects randomly assigned to the stroke self-management intervention to subjects randomly assigned to usual care. Subjects from both groups were assessed at baseline, 3, 6, and 12 months. We delivered the stroke self-management program over 6 months (12 weeks biweekly sessions followed by 12 weeks of bimonthly telephone and group support sessions). Usual care participants received written stroke risk factor materials. The primary outcomes were stroke specific quality of life and the secondary outcomes were stroke self-management, self-efficacy, functioning, and post stroke depression. We are evaluating clinical risk factor management after stroke.

ELIGIBILITY:
Inclusion Criteria:

Patient eligibility criteria include:

* age 18 or older;
* acute diagnosis of ischemic stroke or TIA within past 12 months;
* able to speak and understand English;
* no severe cognitive impairment;
* access to a telephone;
* willing to follow-up in VA/IU Health outpatient care;
* had a previous outpatient primary care visit during the past 12 months in VA/IU Health outpatient care;
* willing to attend all individual phone and group meetings during the 6 month intervention; and
* life expectancy of at least 6 months as defined by the patient's neurologist at stroke event.

Exclusion Criteria:

* Short Portable Mental Status score < 7;
* Significant language comprehension (NIH Stroke Scale commands score > 0); or
* Receptive language deficits (NIH Stroke Scale aphasia score > 2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2013-01-07 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2019-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa M. Damush, PhD, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (2):
- United States (2):
  - Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: Yes
Limited deidentified dataset will be shared after publication completion from study.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Limited de-identified dataset will be shared after publication completion beginning 2022 for 5 years.

REFERENCES:
- [Background] Chen CX, Kroenke K, Stump TE, Kean J, Carpenter JS, Krebs EE, Bair MJ, Damush TM, Monahan PO. Estimating minimally important differences for the PROMIS pain interference scales: results from 3 randomized clinical trials. Pain. 2018 Apr;159(4):775-782. doi: 10.1097/j.pain.0000000000001121. PMID 29200181
- [Result] Chen CX, Kroenke K, Stump T, Kean J, Krebs EE, Bair MJ, Damush T, Monahan PO. Comparative Responsiveness of the PROMIS Pain Interference Short Forms With Legacy Pain Measures: Results From Three Randomized Clinical Trials. J Pain. 2019 Jun;20(6):664-675. doi: 10.1016/j.jpain.2018.11.010. Epub 2018 Dec 6. PMID 30529442
- [Result] Kroenke K, Stump TE, Chen CX, Kean J, Bair MJ, Damush TM, Krebs EE, Monahan PO. Minimally important differences and severity thresholds are estimated for the PROMIS depression scales from three randomized clinical trials. J Affect Disord. 2020 Apr 1;266:100-108. doi: 10.1016/j.jad.2020.01.101. Epub 2020 Jan 23. PMID 32056864
- [Result] Kroenke K, Stump TE, Chen CX, Kean J, Damush TM, Bair MJ, Krebs EE, Monahan PO. Responsiveness of PROMIS and Patient Health Questionnaire (PHQ) Depression Scales in three clinical trials. Health Qual Life Outcomes. 2021 Feb 4;19(1):41. doi: 10.1186/s12955-021-01674-3. PMID 33541362
- [Derived] Kroenke K, Stump TE, Kean J, Krebs EE, Damush TM, Bair MJ, Monahan PO. Diagnostic operating characteristics of PROMIS scales in screening for depression. J Psychosom Res. 2021 Aug;147:110532. doi: 10.1016/j.jpsychores.2021.110532. Epub 2021 May 25. PMID 34052655

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period ran from Jan 7, 2013 through March 31, 2016. Recruitment sites included 2 Veterans Health Administration Medical Facilities, 1 Joint Commission Stroke Center in an urban Hospital, and 1 Safety Net Urban Hospital.
Groups:
- Arm 2 Usual Care: Usual care for treating a patient presenting with an acute ischemic stroke or TIA
Period: Baseline to 6 Month Assessment
Arm/Group | Arm 1 SSM Intervention | Arm 2 Usual Care
Started | 129 | 129
Completed | 113 | 119
Not Completed | 16 | 10
Period: 6 Month to 12 Month Assessment
Arm/Group | Arm 1 SSM Intervention | Arm 2 Usual Care
Started | 113 | 119
Completed | 108 | 116
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- SSM Intervention Arm 1: Stroke self-management program- Participants randomized to this program will receive 6 bi-weekly telephone sessions during the first 3 months followed by 3 monthly reinforcement telephone sessions coupled with 3 monthly group sessions during months 4-6.
  Stroke Self-Management: Stroke self-management program- Participants randomized to this program will receive 6 bi-weekly telephone sessions during the first 3 months followed by 3 monthly reinforcement telephone sessions coupled with 3 monthly group sessions during months 4-6.
- Usual Care Arm 2: Usual care which includes standardized patient education materials on stroke from the American Stroke Association.
- Total: Total of all reporting groups
Arm/Group | SSM Intervention Arm 1 | Usual Care Arm 2 | Total
Number analyzed (Participants) | 129 | 129 | 258
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.09 (10.77) | 62.41 (10.87) | 61.75 (10.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 26 | 49
  Male | 106 | 103 | 209
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 127 | 127 | 254
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 46 | 32 | 78
  White | 77 | 89 | 166
  More than one race | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 129 | 129 | 258
Cerebrovascular Events [Count of Participants; unit: Participants] — Participants who had a diagnosed stroke or TIA as primary diagnoses at discharge from an inpatient admission
  Participants
    Stroke | 109 | 109 | 218
    Transient Ischemic Attack (TIA) | 20 | 20 | 40
National Institute on Health Stroke Scale (NIHSS) [Mean (Standard Deviation); unit: units on a scale] — NIHSS is a clinical assessment of stroke severity and disability at time of stroke. This scale captures total stroke deficits in several domains (consciousness, vision, extraocular movement, facial control, limb strength, ataxia, sensation, and speech and language. Each item is scored and total score is sum of all items. Score ranges from [0 to 42] where 0 reflects no stroke disability and scores between 21-42 indicate severe stroke disability. Scores between 1-4 = minor stroke; Scores between 5-15= moderate stroke; and Scores between 15-20= moderate/severe stroke disability.
  units on a scale | 3.00 (3.20) | 2.96 (2.81) | 2.98 (3.01)
Length of time (days) [Number; unit: Days] — Days from hospital discharge to study enrollment
  Days | 85.74 | 77.20 | 81.47
Stroke Specific Quality of Life [Mean (Standard Deviation); unit: units on a scale] — Stroke Specific, Health-Related Quality of Life. Self-reported measure includes 12 domains over 49 items and an Overall Total Score. Items are scored on a 5 point Likert response format with lower score indicating worse function/lower ability on that item and a higher score indicating better function. Domain score were calculated as an unweighted average of item scores in that specific domain. Overall Stroke Specific, Health-Related Quality of Life = average items 50-62 where a lower score indicates worse health now compared to before the stroke event.
  units on a scale | 3.06 (0.76) | 3.16 (0.73) | 3.11 (0.75)
Self-Efficacy to Manage Stroke Symptoms [Mean (Standard Deviation); unit: units on a scale] — Assesses confidence to manage symptoms and health post stroke on a 1-10 scale where 10 denotes a lot of confidence and 1 denotes no confidence.
  units on a scale | 8.27 (1.72) | 8.47 (1.55) | 8.37 (1.64)

OUTCOME MEASURES:

1. Primary Outcome: Total Stroke Specific Quality of Life
Description: A 49-item instrument that assesses 12 domains relevant to stroke patients' health-related quality of life including: energy, mobility, work, upper extremity function, activities of daily living, family roles, social roles, vision, language, thinking, mood, and personality. A lower score indicates poorer functioning and a higher score indicates better functioning. The minimum value was 1 and maximum value was 5. A Total Stroke Specific Quality of Life Score was calculated as the mean of the 49-items.
Time Frame: Change from baseline to 6 months
Population: Participants were patients discharged with an acute stroke or TIA as the primary diagnoses.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 2 Usual Care: Usual care for acute stroke care services
Arm/Group | Arm 1 SSM Intervention | Arm 2 Usual Care
Number analyzed (Participants) | 129 | 129
units on a scale
  Baseline | 3.80 (0.730) | 3.82 (0.768)
  3 months outcome: number analyzed (Participants) | 116 | 124
  3 months outcome | 4.01 (0.72) | 3.94 (0.79)
  6 months outcome: number analyzed (Participants) | 113 | 119
  6 months outcome | 4.07 (0.75) | 3.95 (0.78)
  Mean Change from 0 to 6 months: number analyzed (Participants) | 113 | 119
  Mean Change from 0 to 6 months | 0.268 (0.06) | 0.133 (0.05)
  Mean Change from 0 to 12 months: number analyzed (Participants) | 108 | 116
  Mean Change from 0 to 12 months | 0.214 (0.04) | 0.181 (0.04)
  12 months outcome: number analyzed (Participants) | 108 | 116
  12 months outcome | 4.02 (0.76) | 4.00 (0.77)
Statistical Analysis 1: Comparison: Arm 1 SSM Intervention vs Arm 2 Usual Care; All the sample size calculations were powered at 80% with a 5% Type I error. We estimated based on our pilot study a change difference of 0.25 on Total Stroke Specific Quality of Life in the intervention group compared to no change in the control group at 6 months. Our power calculations estimated a sample of 226 (113) per group was needed to detect this effect. We used primary outcome row "Mean Change from 0 to 6 months" for this analysis; Test type: Superiority; p = 0.0500, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. Models adjusted for: VA vs Non Va, admission diagnosis (transient ischemic attack vs stroke), sex (male vs female), white vs nonwhite, and baseline total Stroke Specific Quality of life score; Repeated measurements of change GEE analyses of Total Stroke Specific Quality of Life score change at 6 months from baseline; Mean Difference (Net) = 0.14, Standard Error of Mean 0.17 — The adjusted positive mean (standard error) change at 6 months from baseline was higher in the intervention arm compared to in the control arm. Intervention group had 0.14 (SE 0.17) higher improvement compared to the control group
Statistical Analysis 2: Comparison: Arm 1 SSM Intervention vs Arm 2 Usual Care; We evaluated the mean difference on Total Stroke Specific Quality of Life compared to baseline between the intervention and control groups at 12 months using repeated measures ANCOVA models. We used primary outcome row "Mean change from 0 to 12 months" for this analysis; Test type: Superiority; p = 0.26, Mixed Models Analysis — Adjusted least square means (standard errors) adjusted for treatment (Intervention vs control), time of outcome from baseline (3, 6, 12 months), baseline SSQoL, Site (VA vs NonVA), Stroke/TIA diagnosis, sex (m vs f) and race (white vs nonwhite); Mean Difference (Net) = 0.22, Standard Error of Mean 0.04 — Adjusted intervention arm's positive change (regression coefficient with standard error) in Total Stroke Specific Quality of Life was not significantly different at 12 months compared to the control group

ADVERSE EVENTS:
Time Frame: Adverse events were monitored and reported during each assessment period [ 3, 6, and 12 months] after baseline. Participants were asked whether they experienced an adverse or serious adverse event since last contact. If a participant was not available, the interviewer contacted the next of kin listed on the participant contact information provided and asked about adverse events.
Description: All Adverse (AE) and Serious Adverse Events (SAE) and deaths were reported to the Indiana University IRB per protocol. All were reviewed by the IRB and deemed unrelated to our research study.
  SAE were defined as a health event for which the participant was hospitalized for medical care.
  AE were defined as a health event experienced and treated by medical personnel but not hospitalized.
  Deaths were reported as any death occurring during the participant enrollment in the study.
Groups:
- Arm 2 Usual Care: Usual care for acute ischemic stroke
Arm/Group | Arm 1 SSM Intervention | Arm 2 Usual Care
All-Cause Mortality (participants affected / at risk) | 2/129 | 2/129
Serious Adverse Events (participants affected / at risk) | 44/129 | 35/129
Other Adverse Events (participants affected / at risk) | 72/129 | 61/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 SSM Intervention (N=129) | Arm 2 Usual Care (N=129)
CVD related health event (Vascular disorders) | 20 (44) | 8 (35) — Health event required hospitalization
Bone fractures and strains (Musculoskeletal and connective tissue disorders) | 4 (44) | 7 (35) — Falls and injuries
Infection (Infections and infestations) | 5 (44) | 3 (35) — Infections
Kidney stones (Renal and urinary disorders) | 2 (44) | 1 (35)
General disorders (General disorders) | 9 (44) | 13 (35)
Pain (General disorders) | 4 (44) | 3 (35) — Reported pain other than chest pain
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 SSM Intervention (N=129) | Arm 2 Usual Care (N=129)
General Outpatient Care (General disorders) | 72 (72) | 61 (61) — Participant was not hospitalized Any health event for which medical care was received but not admitted into hospital.

LIMITATIONS AND CAVEATS:
Participants who agreed to participate may have had a greater interest in managing their health compared to the general population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2016-05-11): https://cdn.clinicaltrials.gov/large-docs/88/NCT01507688/Prot_SAP_002.pdf
  • Informed Consent Form: Non VA Informed Consent (2016-02-11): https://cdn.clinicaltrials.gov/large-docs/88/NCT01507688/ICF_000.pdf
  • Informed Consent Form: VA Informed consent (2016-02-11): https://cdn.clinicaltrials.gov/large-docs/88/NCT01507688/ICF_001.pdf